CLINICAL TRIAL: NCT05006534
Title: The Efficacy and Adverse Effect of Polatuzumab Vedotin in Patients With Diffuse Large B Cell Lymphoma: an Observation Study
Brief Title: Polatuzumab Vedotin in Patients With Relapsed and Refractory Diffuse Large B Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005095RINA
Record Dates: First submitted 2021-08-01; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Lymphoma
Keywords: Diffuse large B-cell lymphoma; Polatuzumab vedotin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study enrolled patients with relapsed or refractory diffuse large B cell lymphoma treated with polatuzumab vedotin-based chemoimmunotherapies. Patients were allowed to use chemotherapy regimens other than Rituximab and Bendamustine and transplantation following polatuzumab vedotin was also allowed.

DETAILED DESCRIPTION:
Polatuzumab vedotin has been demonstrated to be an effective treatment for patients with relapsed/refractory diffuse large B cell lymphoma in an international phase II clinical trial. The clinical trials was conducted in Europe and the United States. Although there is a phase III trial about polatuzumab vedotin in newly diagnosed patients with diffuse large B cell lymphoma, the double-blind design has limited the efficacy assessment and side effect observation, making it difficult to provide clinicians with further information.

This program hopes to evaluate the clinical course and treatment response of these patients in order to facilitate clinicians' understanding of this drug and to improve patients' quality of life and medical care, as well as to prevent the occurrence of related complications and treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form must be signed before any study specific tests or procedures are done
2. Adult male and female patients ≥20 years at the time of inclusion in the study Ability to understand and follow study-related instructions
3. Histological diagnosis of primary refractory or relapsed aggressive B-cell non-Hodgkin lymphoma (B-NHL), confirmed by a biopsy of involved nodal or extranodal site. Patients with any of the following histologies can be included:

   * DLBCL not otherwise specified (NOS)
   * T-cell/histiocyte-rich large B-cell lymphoma
   * Primary cutaneous DLBCL, leg type
   * Epstein-Barr virus (EBV)-positive DLBCL, NOS
   * DLBCL associated with chronic inflammation
   * Primary mediastinal (thymic) large B-cell lymphoma Refractory disease is defined as no complete remission to first line therapy. Relapsed disease is defined as complete remission to first line therapy followed by disease relapse.
4. Subjects must have received adequate first line therapy including at a minimum: i) anti-CD20 monoclonal antibody unless Investigator determines that tumor is CD20 negative, and ii) an anthracycline containing chemotherapy Regimen
5. Women of childbearing potential must have a negative pregnancy test result within 7 days prior to the first study drug Administration
6. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs
7. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

1. Primary or secondary central nervous system (CNS) lymphoma at the time of recruitment
2. Richter's transformation or prior chronic lymphocytic leukemia (CLL)
3. Vaccination with a live vaccine within 4 weeks prior to Treatment
4. Received polatuzumab vedotin as part of the first line therapy
5. Ongoing treatment or study procedures within any other Investigational Medicinal Product (IMP) clinical trial with the exception of follow-up. In case of a preceding clinical trial, last application of the respective IMP(s) must have been done more than five elimination half-lives before start of study medication in this trial.
6. History of severe allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
7. History of hypersensitivity to any of the study drugs or their ingredients or to drugs with similar structure
8. Pregnancy or breastfeeding, or intending to become pregnant during the study or within 12 months after the last dose of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Polatuzumab vedotin
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival | through study completion, an average of 2 year
  From the use of PoV to death related to any cause

SECONDARY OUTCOMES:
Overall response rate | through study completion, an average of 2 year
  The assessment is based on PET/CT or contrast CT, as determined by the investigator. Including complete remission and partial remission
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 2 year
  Will estimate the safety and tolerability of polatuzumab vedotin when added to intensive chemotherapy regimens

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hong Tsai, MD, MSc, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wang YW, Tsai XC, Hou HA, Tien FM, Liu JH, Chou WC, Ko BS, Chen YW, Lin CC, Cheng CL, Lo MY, Lin YC, Lu LC, Wu SJ, Kuo SH, Hong RL, Huang TC, Yao M. Polatuzumab vedotin-based salvage immunochemotherapy as third-line or beyond treatment for patients with diffuse large B-cell lymphoma: a real-world experience. Ann Hematol. 2022 Feb;101(2):349-358. doi: 10.1007/s00277-021-04711-9. Epub 2021 Nov 11. PMID 34766217